CLINICAL TRIAL: NCT00573482
Title: A Cafeteria Based Study of Weight Gain Prevention
Acronym: Cafeteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Michael R. Lowe, Ph.D., Drexel University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DK02-021 (completed); 5R01HL073775 (NIH)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Obesity; Overweight
Keywords: weight gain prevention; obesity; overweight; food environment; The intervention group received the education in REDE techniques; The control group received no intervention at all.; Both groups were exposed to the food labels and the new lower ED foods.; Only the intervention group received the education sessions and only they were eligible for the price reductions.
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Active Comparator): Control (only exposure to the food labels and the new lower ED foods).
  Interventions: Behavioral: control
- intervention group (Experimental): Education in REDE techniques plus exposure to the food labels and the new lower ED foods.
  Interventions: Behavioral: REDE

INTERVENTIONS:
Behavioral: REDE — The intervention group received the education in REDE techniques.
  The intervention in this study comprised four components:
  * Four group education sessions to introduce the REDE principles of eating;
  * Approximately 10 new lower energy-dense foods were introduced in the employee cafeteria daily at lunchtime;
  * Food labels for all foods sold in the employee cafeteria at lunch time, which provided the energy density, calories, and macronutrient content of the prepared cafeteria foods. Prior to the intervention almost no foods had food labels.
  * Price reductions for lower energy density items. Both groups were exposed to the food labels and the new lower ED foods, but only the intervention group received the education sessions about how to take advantage of the new labels and cafeteria foods and only they were eligible for the price reductions.
  Arms: intervention group
Behavioral: control — The control group received no REDE intervention at all. Both groups were exposed to the food labels and the new lower ED foods, but the control group did not receive the education sessions.
  Arms: control group

SUMMARY:
The dramatic rise in overweight and obesity during the past several decades can be explained by environmental changes that foster increased energy intake and decreased energy expenditure. There are several reasons to suggest that the most effective approach to weight gain prevention is the incorporate reduced-fat eating into an overall strategy of lowering the energy density of the diet. Our energy density manipulations will be designed to reduce both the fat content and the caloric density of foods served at a cafeteria, which serves as the "food environment" for hospital employees.

ELIGIBILITY:
Inclusion Criteria:

* works at one of the two hospitals and eats lunch in the cafeteria 2x per week
* BMI between 23 and 25

Exclusion Criteria:

* current diagnosis of a chronic disease or condition known to affect appetite or body weight
* currently taking medication known to affect appetite or body weight
* current pregnancy or plans to become pregnant within the next 24 months
* current enrollment or plans to enroll within the next 24 months in an organized weight management program
* plans to terminate employment at the hospital within the next 12 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2002-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Weight | 36 months

SECONDARY OUTCOMES:
Caloric and macro-nutrient intake | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lowe, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Local Hospitals, Philadelphia, Pennsylvania, United States